CLINICAL TRIAL: NCT03026998
Title: MRI Screening of Second Primary Cancer Occurring Within Radiation Fields After Treatment by External Beam Radiation Therapy for Hereditary Retinoblastoma
Brief Title: MRI Screening of Second Primary Cancer Occurring Within Radiation Fields After Treatment by External Beam Radiation Therapy for Hereditary Retinoblastoma (DepiSCARRH)
Acronym: DepiSCARRH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IC 2015-14
Record Dates: First submitted 2017-01-06; First posted 2017-01-20 (Estimated); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Hereditary Retinoblastoma
Keywords: hereditary retinoblastoma,; External beam radiation therapy (EBRT)
MeSH Terms: conditions — Retinoblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI (Other)
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — MRI will be performed each year during 10 years.

SUMMARY:
The purpose of this study is to assess the benefit of MR screening for asymptomatic head & neck (or CNS) second primary cancers occurring in hereditary retinoblastoma patients previously treated by external beam radiation therapy (EBRT).

DETAILED DESCRIPTION:
Patients with hereditary retinoblastoma treated during infancy by external beam radiation therapy (EBRT) the risk of second primary cancer occurring within radiation fields is high. The aim of this study is to depict by MRI secondary tumors as early as possible, before the occurrence of clinical symptoms. Affected patients will be further managed in a national expert center with dedicated diagnostic and treatment procedures. However, the benefit of such management has to be assessed in terms of prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Personal history of hereditary retinoblastoma (i.e., familial history of retinoblastoma, or bilateral retinoblastoma, or unilateral multifocal retinoblastoma, or identified germline RB1 mutation or 13q deletion)
* External beam radiation therapy (EBRT) used for retinoblastoma treatment
* Age at inclusion greater or equal to 7 years old.
* Time period between the end of EBRT and inclusion date of 5 years or more
* Written informed consent signed by patient (or legal representative)

Exclusion Criteria:

* Personal history of non-familial unilateral unifocal retinoblastoma without RB1 germline mutation.
* Personal history of second primary neoplasm occurring within radiation fields
* Contraindication for MRI (pacemaker, intraocular metallic foreign body, defibrillators or other implanted electronic devices, intracranial ferro-magnetic clips) or associated conditions preventing from MR examination (intraocular prostheses and implants are not a contraindication for MRI; orthodontic metallic devices are not a contraindication but might decrease the image quality and should be removed, if possible)
* Patients unable to comply with follow-up study requirements, for any geographical, social or psychological reason

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-03-19 (Actual); Primary Completion 2034-03 (Estimated); Study Completion 2034-03 (Estimated)

PRIMARY OUTCOMES:
Assess the benefit of MR screening for asymptomatic head & neck (or CNS) second primary cancers occurring in hereditary retinoblastoma patients previously treated by external beam radiation therapy (EBRT). | Up to 10 years
  Rate of patients with R0-resection quality (versus R1 or R2) among patients with second primary cancer depicted by MRI, with comparison to historical series

SECONDARY OUTCOMES:
Assess the visual prognosis of patients with second primary cancer depicted by MRI | Up to 10 year
  Measure of residual visual functions before and after local treatment of the second primary cancer in patients depicted by MRI compared to that patients who the second primary cancer was depicted by clinical symptoms.
Assess the feasibility of the MR screening program. | Up to 10 years
  Number of MRI performed for the radiological follow-up for patients agreeing to participate to the study.
Number of non tumor detected anomalies with invasive procedures to assess the psychological consequences of the MR screening program | Up to 10 years
Assess the psychological consequences of the MR screening program by the completion of quality of life questionnaires. | Up to 10 years
  - Quality of life questionnaires completed by the patient every year (before MRI) during 10 years.
Number of depicted second primary cancer.to assess the diagnostic accuracy of MRI. | Up to 10 years
Number of asymptomatic depicted second primary cancer by MR to assess the diagnostic accuracy of MRI | Up to 10 years
Number of symptomatic second primary cancer between 2 MRI.to assess the diagnostic accuracy of MRI | Up to 10 years
Measure of sensibility of MRI to detect second primary cancer | Up to 10 years
Measure of specificity of MRI to detect second primary cancer | Up to 10 years
Collection of secondary tumors for future research purpose. | up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Hervé BRISSE, MD, Principal Investigator — NSTITUT CURIE
Locations (1):
- Institut Curie, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).